CLINICAL TRIAL: NCT00974077
Title: Psychophysiological Correlates of Mindfulness and Attention in Recurrent Depression and Healthy Volunteers
Brief Title: Psychophysiological Correlates of Mindfulness Based Cognitive Therapy (MBCT) in Recurrent Depression
Acronym: MBCT & EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Martin Hautzinger, University Professor of Clinical Psychology and Psychotherapy, University Hospital Tuebingen
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HA1399/16-1
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: recurrent depression,; mindfulness training; attention; Evoked EEG potentials; Relapse prevention in recurrent depression
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait List Control (Other): Patients do ot receive psychotherapy. The wait list control group will be assessed according to study protocol and offered MBCT after 6 month
  Interventions: Other: Waiting List Control
- Mindfulness Based Cognitive Therapy (Experimental): The published protocol of MBCT will be used. This is an eight week group program. Participants learn mindfulness techniques but also cognitive techniques to prevent new depressive episodes
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Group treatment over 8 weeks with training in meditation, stress regulation, shift attention, stay present, in addition with cognitive and behavioral strategies (following Williams et al. Manual 2002)
  Arms: Mindfulness Based Cognitive Therapy
Other: Waiting List Control — Patients receive MBCT with a delay of 6 months.
  Arms: Wait List Control

SUMMARY:
The study investigates cognitive attention, rumination and psychophysiological (EEG) processes in healthy subjects and remitted patients with at least three previous depressive episodes. The investigators expect that Mindfulness Based Cognitive Therapy prevents future depressive episodes and has influence on cognitive and psychophysiological measures.

ELIGIBILITY:
Inclusion Criteria:

* recurrent depression with at least 3 previous MD-episodes, currently remitted (no symptoms)

Exclusion Criteria:

* current depression
* lifetime schizophrenia
* bipolar or schizoaffective disorder
* any neurological disorders
* other psychopathology during last 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Relapse (MDE) | 12 month

SECONDARY OUTCOMES:
Electroencephalography (EEG) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hautzinger, PhD, Principal Investigator — Eberhard Karls University
Locations (1):
- Department of Psychology University of Tuebingen, Tübingen, Germany

REFERENCES:
- [Result] Bostanov V, Keune PM, Kotchoubey B, Hautzinger M. Event-related brain potentials reflect increased concentration ability after mindfulness-based cognitive therapy for depression: a randomized clinical trial. Psychiatry Res. 2012 Oct 30;199(3):174-80. doi: 10.1016/j.psychres.2012.05.031. Epub 2012 Jul 6. PMID 22771173
- [Result] Keune PM, Bostanov V, Hautzinger M, Kotchoubey B. Approaching dysphoric mood: state-effects of mindfulness meditation on frontal brain asymmetry. Biol Psychol. 2013 Apr;93(1):105-13. doi: 10.1016/j.biopsycho.2013.01.016. Epub 2013 Feb 11. PMID 23410762